CLINICAL TRIAL: NCT00253487
Title: A Pilot Study of Temozolomide and O-Benzylguanine for Treatment of High-Grade Glioma, Using Autologous Peripheral Blood Stem Cells Genetically Modified for Chemoprotection
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Younger Patients Who Are Undergoing an Autologous Stem Cell Transplant for Newly Diagnosed Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CCHMC-04660; CDR0000446082 (Registry Identifier: PDQ (Physician Data Query)); NCI-7036
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2006-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; childhood high-grade cerebral astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — O(6)-benzylguanine; Busulfan; Temozolomide; Chemotherapy, Adjuvant; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: busulfan
Drug: temozolomide
Procedure: adjuvant therapy
Procedure: autologous bone marrow transplantation
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, busulfan, and O6-benzylguanine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. O6-benzylguanine may also help temozolomide work better by making tumor cells more sensitive to the drug. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy with a peripheral stem cell transplant or bone marrow transplant, using stem cells from the patient that are genetically-modified in the laboratory to protect them from the side effects of chemotherapy, may allow more chemotherapy to be given so that more tumor cells are killed. Giving combination chemotherapy and radiation therapy together with a peripheral stem cell transplant or bone marrow transplant may kill more tumor cells.

PURPOSE: This clinical trial is studying how well giving combination chemotherapy together with radiation therapy works in treating younger patients who are undergoing an autologous stem cell transplant for newly diagnosed gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of a conditioning regimen comprising temozolomide, radiotherapy, and busulfan followed by an infusion of autologous stem cells genetically modified with the MGMT gene and temozolomide and O6-benzylguanine in younger patients with newly diagnosed high-grade gliomas.

Secondary

* Determine the tolerability of intrapatient dose escalation of temozolomide, in terms of transgene expression, in patients treated with this regimen.
* Determine, preliminarily, the antitumor activity of this regimen in these patients.

OUTLINE: This is a pilot study.

* Surgery: Patients undergo biopsy or surgical debulking of the tumor. Two to six weeks later, patients proceed to stem cell mobilization and apheresis.
* Autologous stem cell mobilization and apheresis: Patients receive filgrastim (G-CSF) subcutaneously or IV once daily for at least 4 days before apheresis and continuing until apheresis is complete. Patients undergo apheresis for up to 4 consecutive days until a target number of 5 X 10^6 CD34-positive peripheral blood stem cells (PBSCs) are collected. Patients with insufficient numbers of PBSCs either undergo bone marrow harvest to collect a sufficient number of cells or are removed from the study. The cells are selected for CD34-positive cells which are cryopreserved for later use. Patients then proceed to chemoradiotherapy.
* Chemoradiotherapy: Patients receive oral temozolomide once daily on days 1-42 and undergo radiotherapy once daily, 5 days a week, for 6 weeks. Four to eight weeks later, patients proceed to the low-intensity, nonmyeloablative conditioning regimen.
* Autologous PBSC or bone marrow transduction: Peripheral blood or bone marrow CD34-positive stem cells are transduced with the MGMT gene on day -4.
* Low-intensity, nonmyeloablative conditioning regimen: Patients receive busulfan IV over 2 hours on days -3 and -2. Patients then proceed to autologous PBSC or bone marrow infusion.
* Autologous PBSC or bone marrow infusion: Patients undergo autologous stem cell infusion using transduced PBSCs or bone marrow on day 0. Three to six weeks later, patients proceed to chemotherapy.
* Chemotherapy: Patients receive O6-benzylguanine IV over 1 hour followed by oral temozolomide once daily on days 1-5. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to O6-benzylguanine may receive temozolomide alone. Patients not experiencing dose-limiting toxicity and who have at least 5% transduced neutrophils by peripheral blood analysis after course 1 receive escalating doses (intrapatient) of temozolomide during courses 2-6. Some patients undergo second-look surgery after the first course of chemotherapy.

After completion of study therapy, patients are followed monthly for 3 months, every 3 months for 3 years, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed high-grade glioma of 1 of the following types:

  * Glioblastoma multiforme

    * WHO grade IV disease
  * Anaplastic astrocytoma

    * WHO grade III disease
* No low-grade disease (i.e., WHO grade I-II disease)
* No WHO grade III oligodendroglioma or oligoastrocytoma
* Patients > 30 years of age who have undergone a gross total resection and have nonmeasurable disease as seen on postoperative MRI are eligible
* Measurable disease, as assessed by postoperative MRI, is required in patients ≤ 30 years of age
* No tumor arising in the spine or brainstem
* No metastatic disease in the spine

PATIENT CHARACTERISTICS:

Age

* 5 to 55

Performance status

* Karnofsky 50-100% (for patients 11-30 years of age) OR
* Lansky 50-100% (for patients 5-10 years of age)

Life expectancy

* At least 9 months

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3 (transfusion independent)

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* ALT and AST ≤ 2.5 times upper limit of normal
* Albumin ≥ 2.0 g/dL
* Hepatitis B surface antigen and core antibody negative
* Hepatitis C antibody negative

Renal

* Creatinine normal OR
* Glomerular filtration rate ≥ 70 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Neurologic deficits must be stable or decreasing
* No active infection
* HIV negative
* No other serious illness or medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Concurrent corticosteroids allowed provided dose is stable or decreasing

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Other

* No other concurrent investigational anticancer agents

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2005-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars M. Wagner, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati